CLINICAL TRIAL: NCT07121231
Title: Effectiveness of Motor Support Program in Multidimensional Development of Autistic Children
Brief Title: Motor Support Program for Multidimensional Development in Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülsüm HATİPOĞLU ÖZCAN, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IYYU-KAEK-16-11-2023-01
Record Dates: First submitted 2025-07-23; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Motor support program; Atistic children; Motor skills; Social skills; Pre-academic skills; Sensory motor skills
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: This mixed-method study evaluated the effects of a 12-week Motor Support Program (MSP) on the multidimensional development of children with autism aged 4-6. The program targeted motor skills, social skills, pre-academic abilities, sensory regulation, and autism-specific symptoms. A total of 30 children diagnosed with autism from four special education and rehabilitation centers in Istanbul were randomly assigned to experimental (n = 15) and control (n = 15) groups. Quantitative data were collected using a pretest-posttest control group design: motor skills were measured with BOT-2, social skills with SSRS-PTF, pre-academic skills with PASAF, autism symptoms with the Adapted Autism Behavior Checklist, and sensory processing with the Sensory Profile. Qualitative data were obtained through semi-structured focus group interviews with parents, each lasting approximately 30 minutes. The interview questions were developed by the researchers and finalized based on expert feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Support Program (Experimental): Participants in this group completed a motor skills support program designed with a holistic approach to support cognitive development through concepts such as color, shape, and number, as well as social skills such as greeting, lining up, and cooperation, through activities based on basic motor skills such as throwing, catching, running, and jumping.
  Interventions: Other: Motor Support Program
- Standard Education (No Motor Support) (No Intervention): Participants in the control group continued their individual education programs. However, they did not participate in any physiotherapy or motor support programs. Only pre- and post-test measurements were taken.

INTERVENTIONS:
Other: Motor Support Program — The MSP was implemented over 12 weeks, two days a week, 50 minutes per session. Based on pre-test results, 30% (15 minutes) of each session was devoted to individualized activities, and 70% (35 minutes) to group activities supporting peer interaction. This structure allowed for both personalized support and social engagement. The program was carried out by the research team and eight special education teachers at the children's rehabilitation centers. Each child received one-on-one support from at least one teacher. Activities were aligned with preschool motor development goals and followed a four-phase structure: (1) Warm-up (5 min): rhythmic movements (e.g., walking, running, jumping); (2) Preparation (5 min): functional exercises for flexibility and joint mobility; (3) Main activity (35 min): individual and group exercises to enhance motor, social, and pre-academic skills; (4) Cool-down (5 min): group games reinforcing learned skills and social interaction.
  Arms: Motor Support Program

SUMMARY:
This mixed-method study evaluated the effects of a 12-week Motor Support Program (MSP) on the multidimensional development of children with autism aged 4-6. The program targeted motor skills, social skills, pre-academic abilities, sensory regulation, and autism-specific symptoms. A total of 30 children diagnosed with autism from four special education and rehabilitation centers in Istanbul were randomly assigned to experimental (n = 15) and control (n = 15) groups. Quantitative data were collected using a pretest-posttest control group design: motor skills were measured with BOT-2, social skills with SSRS-PTF, pre-academic skills with PASAF, autism symptoms with the Adapted Autism Behavior Checklist, and sensory processing with the Sensory Profile. Qualitative data were obtained through semi-structured focus group interviews with parents, each lasting approximately 30 minutes. The interview questions were developed by the researchers and finalized based on expert feedback.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of the Motor Support Program applied to autistic children aged 4-6 years on motor skills, social skills, pre-academic skills, sensory regulation and autism-specific symptoms from a multidimensional and holistic perspective. In this respect, the study aims to contribute to the limited literature on the subject by addressing these developmental areas within the same intervention program and to provide a scientific basis for the planning of motor support programs as an alternative application in preschool education programs for autistic children.

This study was designed with a mixed method approach. Mixed method is an approach that aims to address research problems in a more in-depth and multidimensional way by combining the strengths of quantitative and qualitative research traditions. In the quantitative dimension of the study, the effects of the motor support program (MSP) applied to children with autism on motor skills, social skills, pre-academic skills, sensory profile and autism symptoms were evaluated with a pretest-posttest control group design. Qualitative data were collected through focus group interviews with parents, and family observations were analyzed in accordance with Braun and Clarke's (2006) thematic analysis process. Interviews were analyzed with open codes and themes were created according to content similarities.

The participants of the study consisted of a total of 30 children between the ages of 4-6 years diagnosed with autism attending four different special education and rehabilitation centers in Istanbul. This number of participants, determined as a result of the G*Power analysis, was assigned equally to the experimental (n = 15) and control (n = 15) groups by random number generation method using Excel software. All participants were included in the study with the written consent of their parents, who were informed about the conditions of participation in the study. The inclusion criteria were that the participants were between the ages of 4 and 6, had been diagnosed with autism, had not participated in any MSP before, did not have a health problem that would constitute an obstacle to MSP implementation, and did not have secondary diagnoses such as visual or hearing impairment. The exclusion criteria included the detection of a health problem that prevented children in the experimental group from participating in the MSP, the participants in the experimental or control group not participating in the assessment tests, or voluntarily leaving the training or measurement process.

The Bruininks-Oseretsky Motor Competence Test-2 (BOT-2) was used to assess motor skills and took approximately 10-15 minutes for each child. The Pre-Academic Skills Assessment Form (PASAF), which was used to measure pre-academic skills, was administered in approximately 10-15 minutes. In the assessment of social skills, the Social Skills Assessment System Preschool Teacher Form (SSRS-PTF) was completed by the children's special education teachers in approximately 10 minutes for each child. The Adapted Autism Behavior Checklist, which was administered through face-to-face interviews with parents to determine the level of autism symptoms, took approximately 25-30 minutes for each child. Also, the interview questions used for the qualitative component were developed by the researchers and finalized following expert review. The data were collected through semi-structured interviews lasting approximately 30 minutes.

During the teaching sessions of the MSP in the implementation process, teaching strategies that are sensitive to the learning needs of autistic children were used. Pedagogical approaches such as structured instruction supported by activity charts and visual cues, guidance with clear and short instructions, allowing the child to make choices, providing concrete experiences and modeling were taken as basis. In this way, progress was made in the teaching process of each skill area with methods that were sensitive to individual differences and proven to be effective. At the end of each session, the child's interest and performance in the activities were evaluated with observation forms and these evaluations formed the basis for planning the next training sessions.The program was implemented by the researchers in the special education and rehabilitation centers where the children were studying. The implementation process lasted a total of 12 weeks, two days a week, 50 minutes a day. In line with the pre-test results, 30% (15 minutes) of the sessions were allocated to individual activities and 70% (35 minutes) to group activities that enabled children to interact, taking into account the areas that each child needed to be supported individually. Thus, in each session, both individualized support was provided and group activities that emphasized social interaction were intensively implemented. MSP implementations were carried out in the presence of the research team and eight special education teachers working in the institutions where the children attended. Each child was individually supported by at least one special education teacher during the implementation.The activities were structured in line with the motor development goals and physical activity outcomes of the preschool period. The implementation sessions have a four-stage structure: Warm-up phase: Consists of rhythmic warm-up movements such as walking, running, jumping (5 minutes); Preparation phase: Physical preparation for the target skills is provided with functional exercises that improve joint mobility and flexibility (5 minutes); Main activity phase: Consists of individual and group activities based on basic movement skills, supporting motor, social and pre-academic skills (35 minutes); and End phase: The session ends with games played with the participation of the whole group, reinforcing target skills and increasing social interaction (5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Participants were between the ages of 4 and 6.
* Had been diagnosed with autism.
* Had not participated in any Motor Skills Program (MSP) before.
* Did not have any health problems that would prevent MSP implementation.
* Did not have secondary diagnoses, such as visual or hearing impairment.

Exclusion Criteria:

* Detection of a health problem that prevented children in the experimental group from participating in the MSP.
* Non-participation in the assessment tests by participants in either the experimental or control group.
* Voluntary withdrawal from the training or measurement process.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Change in Social Skills as Measured by the Social Skills Assessment System - Preschool Teacher Form (SSRS-PTF) | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest), and 12 weeks after the completion of the intervention (follow-up test).
  This scale is a behavioral assessment tool that can be applied to children aged 3-18. The form, which is structured for the preschool period, consists of a total of 40 items and two subscales. The first 30 items assess social skills such as cooperation, taking responsibility, and self-regulation, while items 31-40 measure problem behaviors such as aggression, stubbornness, and noncompliance with rules. The scale is evaluated using a three-point Likert-type scoring system for each item: "never" (0), 'sometimes' (1), and "very often" (2). The maximum score that can be obtained on the Social Skills subscale is 90, with higher scores indicating more developed social skills in the child. The maximum score that can be obtained on the Problem Behaviors subscale is 30, and a score closer to zero indicates that problem behaviors are less frequent.
Change in Motor Skills as Measured by the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition - Short Form (BOT-2 SF)" | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest), and 12 weeks after the completion of the intervention (follow-up test).
  In this study, the short form of the Bruininks-Oseretsky Motor Competence Test-2 (BOT-2 SF), which was developed to assess the motor skill levels of individuals aged 4-21 years, was used. The short form used in the study consists of a total of eight subtests and 12 items. These subtests include fine motor accuracy, fine motor integration, manual agility, two-way coordination, balance, running speed and agility, hand-arm coordination and strength. The maximum score that can be obtained in the test is 50. As the total score increases, the level of motor skills increases.
Change in Pre-Academic Skills as measured by Pre-Academic Skills Assessment Form | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest), and 12 weeks after the completion of the intervention (follow-up test).
  The Pre-Academic Skills Assessment Form (PASAF) developed by Özcan (2022) is an assessment form that can be applied to typically developing children and children with special needs between the ages of 3 and 6. The basic concepts determined in line with the goals of preschool education are grouped under the headings of color, geometric shape, size and number, and the form consists of 4 subtests and a total of 34 items. The scoring criteria of PASAF are based on scoring each item as 1 (one) or 0 (zero). A score of 1 indicates that the child responded correctly to the relevant item, while a score of 0 indicates that the child responded incorrectly or did not respond. As the total score increases, the level of prior academic skills improves.

SECONDARY OUTCOMES:
Adapted Autism Behavior Checklist to assess symptoms related to autism | Evaluations were conducted at two time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  The Adapted Autism Behavior Checklist (A-ABC), first published by Krug, Arick, and Almond in 1980, is based on the Autism Behavior Checklist (ABC) [53]. In Turkey, this measurement tool was structured within the Autism Spectrum Disorder Comprehensive Assessment Set (IVO-ODS) and adapted by Özdemir and colleagues (2013). The validity and reliability analyses of the Turkish version of the scale were conducted by Özdemir (2014) [55]. A-ABC is a structured observation tool that aims to systematically assess the behavioral patterns of children with autism and determine the level of support needed by the individual. The scale provides information in basic areas such as communication, social interaction, sensory reactions and problem behaviors. As a result of the assessment, children's support needs are classified as mild, moderate or high.
Sensory profile questionnaire to assess sensory motor skills | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest), and 12 weeks after the completion of the intervention (follow-up test).
  The Sensory Profile Scala was designed by Dunn in 1999 to assess children's sensory processing skills and is administered to children aged 3-10 years [58]. The scale aims to assess the sensory reactions of children in their daily lives and is completed by the caregiver. Turkish adaptation, validity and reliability study was conducted by Kayıhan et al. The Sensory Profile Scale consists of three main sections and their sub-sections: (1) Sensory processing, (2) Sensory modulation, and (3) Behavioral-emotional responses. The scale, which consists of 125 items in total, is structured to assess the frequency of children's behaviors in response to different sensory stimuli. The items are scored on a 5-point Likert-type rating system. In this system, "Always" response is evaluated as 1 point and "Never" response is evaluated as 5 points.As the total score on the scale increases, sensory regulation skills improve.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aykır A, Tekinarslan İ. C. Adaptation of the Social Skills Rating System (SBDS) preschool teacher form into Turkish: A validity and reliability study. Education and Science. 2012; 37(165): 3-17.
- [Background] Kayıhan H, Günel M. K, Bumin G. Adaptation of the Sensory Profile into Turkish for children aged 3-10 years: A validity and reliability study. Turkish Journal of Physiotherapy and Rehabilitation. 2011; 22(2): 44-53.
- [Background] Özcan G. H. Otizm Spektrum Bozukluğu Tanısı Almış Çocuklarda Hareket Eğitimi Programının Akademik Beceriler, Motor Beceriler ve Sosyal İletişim Becerileri Üzerindeki Etkisinin İncelenmesi (PhD thesis) İstanbul: Marmara University; 2022.
- [Background] Krug DA, Arick J, Almond P. Behavior checklist for identifying severely handicapped individuals with high levels of autistic behavior. J Child Psychol Psychiatry. 1980 Jul;21(3):221-9. doi: 10.1111/j.1469-7610.1980.tb01797.x. No abstract available. PMID 7430288